CLINICAL TRIAL: NCT06922812
Title: Intermittent White Light Stimulation (IWLS) for the Treatment of Major Depressive Disorder: An Open-Label Pilot Study of Safety, Tolerability, and Preliminary Efficacy
Brief Title: IWLS for Major Depressive Disorder: An Open-Label Study of Safety, Tolerability, and Efficacy
Acronym: IWLS-MDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre R Brunoni, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 84990324.7.0000.0068
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: open-label clinical trial; light; 60 Hz; major depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IWLS Intervention (Experimental): Participants in this arm will receive Intermittent White Light Stimulation (IWLS) at 60 Hz using an LED-equipped eye mask. Sessions will occur once daily (Monday to Friday) for 2 consecutive weeks, totaling 10 sessions. Each session will last 30 minutes. Follow-up assessments will be conducted at weeks 4 and 6 after the intervention period. The device used is developed by SyntropicMedical (Austria) and emits approximately 700 lux of diffuse white light delivered tangentially to the eyes.
  Interventions: Device: Intermittent White Light Stimulation (IWLS)

INTERVENTIONS:
Device: Intermittent White Light Stimulation (IWLS) — A wearable device developed by SyntropicMedical (Austria) delivers intermittent white light at 60 Hz using LED strips embedded in safety goggles. The light is diffused (approximately 700 lux) and projected tangentially to the participant's eyes. Participants will undergo 10 daily sessions (30 minutes each) over a two-week period. The intervention aims to evaluate the safety, tolerability, and potential antidepressant effects of 60 Hz visual stimulation in individuals with moderate to severe Major Depressive Disorder.

SUMMARY:
INTRODUCTION:

Depression is the most common mood disorder worldwide, with approximately 20 million adults affected in the United States in 2019. Current pharmacological treatments are not effective for all patients, often have significant side effects, and in some cases, require medical monitoring. Non-invasive brain stimulation (NIBS) techniques are emerging as a promising therapeutic alternative, offering fewer side effects. In this context, 60 Hz intermittent light stimulation may represent a promising and safe treatment option for depression. Animal studies have demonstrated that this form of stimulation can promote neuroplasticity, while studies in healthy individuals have shown the technique to be safe. However, 60 Hz intermittent light stimulation has not yet been evaluated in depressed patients in clinical trials.

METHODS:

This is an open-label study designed to assess the safety and tolerability of 60 Hz intermittent light stimulation (ILS) in individuals with moderate to severe depression. The trial will last six weeks in total, consisting of five sessions per week during the first two weeks, with one daily session (a total of 10 sessions, each lasting 30 minutes with 60 Hz white light stimulation), followed by two follow-up visits at weeks 4 and 6. Thirty patients aged 18 to 59 years with a current diagnosis of moderate to severe major depressive episode (HDRS-17 > 16) and a stable antidepressant regimen for at least six weeks will be recruited. The primary outcome will be the safety and tolerability of the device. Clinical improvement will be assessed through changes in HDRS-17 scores and other validated depression and anxiety scales.

EXPECTED RESULTS:

The results of this pilot study may advance knowledge in the field and pave the way for future placebo-controlled clinical trials.

DETAILED DESCRIPTION:
This is an open-label pilot study evaluating the safety, tolerability, and preliminary efficacy of Intermittent White Light Stimulation (IWLS) in individuals with moderate to severe Major Depressive Disorder. The intervention consists of 10 sessions over two weeks, with follow-up at weeks 4 and 6. The study aims to gather data to support future randomized controlled trials using IWLS for depression.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Current diagnosis of Major Depressive Disorder (MDD), confirmed by MINI;
* HDRS-17 score ≥16 at baseline;
* Stable antidepressant regimen for at least 6 weeks prior to enrollment;
* Able and willing to provide informed consent.

Exclusion Criteria:

* Diagnosis of other psychiatric disorders (e.g., bipolar disorder, psychotic disorders, OCD, ADHD, personality disorders, dementia);
* Substance or alcohol use disorders;
* Severe suicidal ideation or psychotic symptoms;
* HDRS-17 score >28;
* Neurological or severe medical conditions;
* History of epilepsy, migraine, or photosensitivity;
* Retinal disease or cataracts;
* Regular use of anti-inflammatory medications or clopidogrel;
* Any worsening of symptoms during the trial (e.g., psychosis, HDRS >28, or suicidal ideation);
* Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of Intermittent White Light Stimulation (IWLS) | 6 weeks
  Safety and tolerability will be assessed through adverse events reported by participants during the stimulation period and follow-up, as well as dropout rates. Adverse effects such as dry eyes, headache, drowsiness, or discomfort will be recorded using a structured questionnaire. Ophthalmologic examinations will be conducted at baseline and at 6 weeks.

SECONDARY OUTCOMES:
Change in Depression Severity as Measured by HDRS-17 | Baseline, Day 12, Day 40
  Depressive symptoms will be evaluated using the 17-item Hamilton Depression Rating Scale (HDRS-17). Outcomes will include change from baseline, clinical response (≥50% reduction), and remission (score <7) at Days 12 and 40.

CONTACTS AND LOCATIONS:
Overall Officials: Kallene Vidal, Doctor, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided